CLINICAL TRIAL: NCT00511108
Title: A Phase I Double-Blind, Randomized, Placebo-Controlled Clinical Trial to Study the Safety, Efficacy, and Mechanism of Action of Sitagliptin and Pioglitazone in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Diet and Exercise
Brief Title: Sitagliptin and Pioglitazone Mechanism of Action Study in Type 2 Diabetes Mellitus (0431-061)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-061; MK0431-061; 2007_530
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Results first posted 2010-03-05 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): Arm 1: drug
  Interventions: Drug: Comparator: sitagliptin phosphate; Drug: Comparator: placebo to pioglitazone
- 2 (Active Comparator): Arm 2: active comparator
  Interventions: Drug: Comparator: pioglitazone; Drug: Comparator: placebo to sitagliptin
- 3 (Experimental): Arm 3: drug + active comparator
  Interventions: Drug: Comparator: sitagliptin phosphate; Drug: Comparator: pioglitazone
- 4 (Placebo Comparator): Arm 4: placebo comparator
  Interventions: Drug: Comparator: placebo to pioglitazone; Drug: Comparator: placebo to sitagliptin

INTERVENTIONS:
Drug: Comparator: sitagliptin phosphate — sitagliptin phosphate 100 mg as oral tablets. Each patient will be administered 1 tablet once daily.
  Arms: 1; 3
Drug: Comparator: pioglitazone — pioglitazone 30 mg will be supplied as oral tablets. Each patient will be administered 1 tablet once daily.
  Arms: 2; 3
Drug: Comparator: placebo to pioglitazone — pioglitazone 30 mg placebos will be supplied as oral tablets. Each patient will be administered 1 tablet once daily.
  Arms: 1; 4
Drug: Comparator: placebo to sitagliptin — sitagliptin phosphate 100 mg placebos will be supplied as oral tablets. Each patient will be administered 1 tablet once daily.
  Arms: 2; 4

SUMMARY:
A clinical study to determine the safety, efficacy and mechanism of action of sitagliptin alone and in combination with pioglitazone, in patients with type 2 diabetes mellitus who have inadequate glycemic (blood sugar) control.

ELIGIBILITY:
Inclusion Criteria:

* Patient has type 2 diabetes mellitus
* Male
* Female that is highly unlikely to become pregnant
* Patient is not on an antihyperglycemic agent (AHA) (hemoglobin A1c [A1C] 7-10%) or on oral single AHA or low-dose combination therapy (A1C 6.5-9.0%)

Exclusion Criteria:

* Patient has a history of type 1 diabetes mellitus or a history of ketoacidosis
* Patient has required insulin therapy within the past 12 weeks
* Patient is on or has been taking a Peroxisome Proliferator-Activated Receptor-gamma (PPAR -gamma) agent (i.e. Thiazolidinediones [TZDs]) within the prior 12 weeks of the screening visit.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2007-07-11 (Actual); Primary Completion 2009-02-24 (Actual); Study Completion 2009-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Alba M, Ahren B, Inzucchi SE, Guan Y, Mallick M, Xu L, O'Neill EA, Williams-Herman DE, Kaufman KD, Goldstein BJ. Sitagliptin and pioglitazone provide complementary effects on postprandial glucose and pancreatic islet cell function. Diabetes Obes Metab. 2013 Dec;15(12):1101-10. doi: 10.1111/dom.12145. Epub 2013 Jul 19. PMID 23782502

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 12-Sep-2007; Last Patient Last Visit: 24-Feb-2009
  Forty-four medical clinics worldwide (17 in the United States, 20 in Europe, 4 in Australia, and 3 in Israel).
Pre-assignment Details: Patients 30-65 years of age with type 2 diabetes mellitus (T2DM) with inadequate glycemic control (fasting plasma glucose [FPG] 130-260 mg/dL [7.2-14.4 mmol/L]) on diet and exercise alone were eligible for randomization.
Groups:
- Sitagliptin 100 mg: Includes patients receiving once-daily administration of sitagliptin 100 mg and matching placebo to pioglitazone 30 mg.
- Pioglitazone 30 mg: Includes patients receiving once-daily administration of pioglitazone 30 mg and matching placebo to sitagliptin 100 mg.
- Sitagliptin 100 mg + Pioglitazone 30 mg: Includes patients receiving once-daily administration of sitagliptin 100 mg and pioglitazone 30 mg.
- Placebo: Includes patients receiving once-daily administration of matching placebo to sitagliptin 100 mg and matching placebo to pioglitazone 30 mg.
Period: Overall Study
Arm/Group | Sitagliptin 100 mg | Pioglitazone 30 mg | Sitagliptin 100 mg + Pioglitazone 30 mg | Placebo
Started | 52 | 54 | 52 | 53
Completed | 46 | 52 | 47 | 48
Not Completed | 6 | 2 | 5 | 5
Not completed — Adverse Event | 2 | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg | Pioglitazone 30 mg | Sitagliptin 100 mg + Pioglitazone 30 mg | Placebo | Total
Number analyzed (Participants) | 52 | 54 | 52 | 53 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (7.6) | 53.4 (7.8) | 53.3 (8.6) | 53.3 (7.7) | 53.6 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 31 | 18 | 21 | 94
  Male | 28 | 23 | 34 | 32 | 117
Race/Ethnicity, Customized [Number; unit: participants]
  White | 45 | 43 | 49 | 48 | 185
  Black | 6 | 9 | 3 | 2 | 20
  Asian | 1 | 1 | 0 | 2 | 4
  Other | 0 | 1 | 0 | 1 | 2
Glucose 5-hour (hr) Total area under the curve (AUC) [Mean (Standard Deviation); unit: mg*hr/dL] — Glucose concentration was measured at 11 points during a Meal Tolerance Test (MTT), at times -10, 0, 10, 20, 30, 60, 90, 120, 180, 240, 300 minutes. Total AUC was calculated over 5 hours including all sample points starting from 0 minutes using the trapezoid method.
  The number of participants for the "Sitagliptin 100 mg + Pioglitazone 30 mg" arm is 51, making the total number of participants for this measure 210.
  mg*hr/dL | 1179.9 (322.8) | 1250.6 (349.6) | 1276.0 (348.5) | 1255.1 (290.9) | 1240.4 (328.4)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent] | 7.7 (0.8) | 7.9 (0.9) | 7.9 (0.9) | 8.0 (1.1) | 7.9 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glucagon 3-hour Total Area Under the Curve (AUC) After 12 Weeks of Treatment
Description: Glucagon concentration was measured at 9 points during an Meal Tolerance Test (MTT), at times -10, 0, 10, 20, 30, 60, 90, 120, and 180 minutes. Total AUC was calculated over 3 hours including all sample points starting from 0 minutes using the trapezoid method. The change from baseline reflects Week 12 total AUC minus the Week 0 total AUC.
Time Frame: Baseline and 12 weeks
Population: The Full Analysis Set (FAS) included all patients with a baseline value and ≥1 post-baseline value for this outcome. For FAS patients with no data at Week 12, the last observed measurement was carried forward to Week 12.
Measure: Least Squares Mean (95% Confidence Interval); unit: pg*hr/mL
Arm/Group | Sitagliptin 100 mg | Pioglitazone 30 mg | Sitagliptin 100 mg + Pioglitazone 30 mg | Placebo
Number analyzed (Participants) | 48 | 47 | 42 | 39
pg*hr/mL | -17.2 [-30.1 to -4.2] | -4.9 [-18.1 to 8.3] | -29.8 [-43.6 to -16.1] | 12.5 [-1.9 to 26.9]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA; Model terms: treatment, prior diabetes pharmacotherapy (yes or no), and baseline value as a covariate; Mean Difference (Net) = -29.7, 95% CI [-48.7 to -10.6]

2. Primary Outcome: Percent Change From Baseline in Index of Static Beta-cell Sensitivity to Glucose After 12 Weeks of Treatment
Description: Static sensitivity is a measure of the effect of glucose on beta cell secretion and is the ratio between the insulin secretion rate and glucose concentration above the threshold level at steady state.
  Percent change from baseline was calculated as the difference between index of static sensitivities at Week 12 and at baseline with respect to the index of static sensitivity at baseline times 100.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Sitagliptin 100 mg | Pioglitazone 30 mg | Sitagliptin 100 mg + Pioglitazone 30 mg | Placebo
Number analyzed (Participants) | 38 | 34 | 27 | 33
Percent Change | 71.5 [46.8 to 100.3] | 27.0 [7.8 to 49.7] | 125.2 [87.2 to 171.0] | -2.3 [-17.4 to 15.5]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, prior diabetes pharmacotherapy (yes or no), and log-scaled baseline value as a covariate; Geometric Mean Difference = 73.8, 95% CI [44.2 to 104.4] — The outcome was analyzed by ANCOVA on the log scale. Results have been back-transformed to the original scale

3. Secondary Outcome: Change From Baseline in Glucose 5-hour Total AUC After 12 Weeks of Treatment
Description: Glucose concentration was measured at 11 points during an Meal Tolerance Test (MTT), at times -10, 0, 10, 20, 30, 60, 90, 120, 180, 240, 300 minutes. Total AUC was calculated over 5 hours including all sample points starting from 0 minutes using the trapezoid method. The change from baseline reflects Week 12 total AUC minus the Week 0 total AUC.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg*hr/dL
Arm/Group | Sitagliptin 100 mg | Pioglitazone 30 mg | Sitagliptin 100 mg + Pioglitazone 30 mg | Placebo
Number analyzed (Participants) | 48 | 49 | 44 | 42
mg*hr/dL | -209.8 [-281.6 to -138.0] | -245.6 [-316.6 to -174.6] | -389.2 [-463.6 to -314.7] | 18.6 [-58.2 to 95.4]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg + Pioglitazone 30 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, prior diabetes pharmacotherapy (yes or no), and baseline value as a covariate; Mean Difference (Net) = -407.8, 95% CI [-513.4 to -302.1]

ADVERSE EVENTS:
Time Frame: Weeks 0-12
Arm/Group | Sitagliptin 100 mg | Pioglitazone 30 mg | Sitagliptin 100 mg + Pioglitazone 30 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/52 | 0/54 | 1/52 | 0/53
Other Adverse Events (participants affected / at risk) | 3/52 | 3/54 | 0/52 | 9/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg (N=52) | Pioglitazone 30 mg (N=54) | Sitagliptin 100 mg + Pioglitazone 30 mg (N=52) | Placebo (N=53)
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg (N=52) | Pioglitazone 30 mg (N=54) | Sitagliptin 100 mg + Pioglitazone 30 mg (N=52) | Placebo (N=53)
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 0 | 3
Blood glucose increased (Investigations) | 0 | 0 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.